CLINICAL TRIAL: NCT02513849
Title: A Pilot Study of Tamoxifen in Oesophageal Cancer
Brief Title: Tamoxifen in Patients With Oesophageal Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 15021; 163909 (Registry Identifier: IRAS)
Record Dates: First submitted 2015-07-22; First posted 2015-08-03 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Cancer; Gastrointestinal Neoplasms
Keywords: esophagus; gastroscopy; tamoxifen
MeSH Terms: conditions — Neoplasms; Gastrointestinal Neoplasms | interventions — Tamoxifen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tamoxifen treatment (Experimental): Patients will be administered tamoxifen, 80mg/ day orally for 4 days as a loading dose, followed by 20mg/ day thereafter until gastroscopy and biopsy 4 weeks later.
  Interventions: Drug: Tamoxifen

INTERVENTIONS:
Drug: Tamoxifen — Daily tamoxifen tablet for approximately 4 weeks
  Other Names: Tamoxifen Citrate

SUMMARY:
Cancer of the gullet (oesophagus) is a lethal disease in which only 15% of patients survive 5 years once diagnosed. It is more common in men than women, and men appear to have a worse prognosis. One suggestion for this gender difference is the sex hormone oestrogen, which exerts its effect via oestrogen receptors. The role of oestrogen in breast cancer is well described, and antioestrogen medication such as tamoxifen, which blocks oestrogen receptors are in widespread and effective use. The role of oestrogen receptors in oesophageal cancer however, is less well defined. Work conducted by the investigators, as well as another research group in Australia showed that antioestrogens including tamoxifen, reduce oesophageal cancer cell growth in the laboratory. To date, no studies have assessed the effect of tamoxifen therapy on oesophageal cancer growth in humans. The investigators propose a study to determine the effect of tamoxifen in patients with oesophageal cancer who aren't undergoing surgery or chemotherapy. Patients will receive tamoxifen tablets daily for 4 weeks after which time a biopsy (sample of cancer tissue) will be taken at gastroscopy (a flexible camera that is passed into the mouth through the gullet into the stomach). The biopsy will be compared with the biopsy taken at the time of diagnosis to determine if tamoxifen has had any effect on cancer cell growth. If this study shows that tamoxifen does slow cancer cell growth it could lead to a larger study of patients with oesophageal cancer taking tamoxifen for a longer time period to determine if there is any clinical benefit.

DETAILED DESCRIPTION:
Oesophageal cancer is the eighth most common cancer worldwide, and the United Kingdom (UK), has the world's highest incidence of oesophageal adenocarcinoma. The 5- year survival for patients diagnosed with oesophageal cancer during 2010-2011 in England and Wales was 15%. Ten- year survival for oesophageal cancer in the UK ranks the third lowest out of 20 common cancers, and only one-third of patients are candidates for surgical resection at presentation. Interestingly, oesophageal cancer is a male dominant disease with a male: female ratio of 5:1 to 10:1. Most published epidemiological evidence has been unable to find any differences in exposure to known risk factors of oesophageal cancer between the two genders, and it has been suggested that oestrogen, which exerts its effect via oestrogen receptors, could be responsible for the gender bias.

Recent work from the investigators Academic Unit (Faculty of Medicine and Health Sciences, University of Nottingham, Royal Derby Hospital, Derby), found increased expression of oestrogen receptors in oesophageal cancer compared to matched normal mucosal samples, and up-regulation of oestrogen receptors was associated with poor survival outcomes. This association between oestrogen receptor expression and oesophageal cancer has also been demonstrated in numerous other studies. The investigators research also showed that blocking oestrogen receptors using highly selective antagonists (MPP and PHTPP) or the selective oestrogen receptor modulators, tamoxifen and raloxifene significantly inhibited oesophageal cancer cell proliferation in vitro (p <0.05). Similar findings have been found by another research group using tamoxifen and raloxifene. To date, there are no published studies assessing the effect of tamoxifen in patients with oesophageal adenocarcinoma in vivo. The investigators propose an initial pilot study to determine the effects of short-term tamoxifen on biological parameters in oesophageal cancer. Determination of any biological response will potentially allow for a further phase I study to determine any clinical response.

The biological response to treatment will be assessed by immunohistochemistry using a monoclonal antibody to Ki67, a nuclear antigen present throughout the cell cycle (GI, S, G2 and M phases) of proliferating cells but absent in quiescent (GO) cells. The percentage change of Ki67 expression in the oesophageal cancer biopsy tissue taken at diagnosis (pre- tamoxifen), with the paired biopsy taken after 4 weeks of tamoxifen will provide information the antitumor effect of tamoxifen on oesophageal cancer. Ki67 expression has been used as a biomarker of tamoxifen therapy in numerous breast cancer studies on matched breast core biopsy specimens or fine needle aspiration cytology specimens 20-36. Of the studies reviewed, all reported a decrease in Ki67 expression, which was significant in 10 out of 18 studies after a median of 28 days (range: 14 - 84 days) of 20mg/ day of tamoxifen, in a median of 51 patients (10 - 201 patients). The use of Ki67 as a biomarker of tamoxifen therapy has also been used in a study of 24 patients with cervical cancer who received 80mg tamoxifen for 5 days. The study reported a drop in the median Ki67 Labelling Index from 5.6% in the pre- tamoxifen biopsy tissue to 3.0% post- tamoxifen (P < 0.001). The cervical cancer biopsy samples used are similar in size to the oesophageal biopsies we will be using in this study, and we are confident a measure of Ki67 expression is the most suitable biomarker available to assess the biological response to tamoxifen.

Tamoxifen has been the gold standard endocrine treatment for oestrogen receptor positive breast cancer for over 30 years, following FDA-approval by the US Food and Drug Administration in 1977. It is estimated that more than 400,000 women are alive today as a result of tamoxifen, and millions more have benefited from palliation and extended disease-free survival. It was initially licensed for use in metastatic disease, followed by use in the adjuvant setting, and has recently been commissioned for breast cancer chemoprevention by the National Institute for Health and Care Excellence. A meta-analyses of 20 trials showed tamoxifen treatment was associated with a reduction in disease recurrence by 39%, and mortality by 30%. The hope is that patients with oesophageal cancer treated with tamoxifen would have improved clinical outcomes similar to those observed in patients with breast cancer. To observe such a clinical benefit patients would have to take tamoxifen for an extended period of time like in breast cancer, where in the adjuvant setting, treatment is for 5 years, which may be increased to 10 years for even further clinical benefit according to evidence reported in two recent phase III trials. Currently, there is not enough evidence available to justify a study of long-term tamoxifen in patients with oesophageal cancer, and so this initial pilot study is to determine any biological response of oesophageal cancer to short-term tamoxifen.

Despite its widespread use, the optimal in vivo therapeutic concentration range for tamoxifen remains to be established because of a lack of dose-response studies, and a high degree of inter-individual variability in steady-state levels of tamoxifen and its metabolites. Patients enrolled in this study will receive 80mg of tamoxifen for the first 4 days followed by 20mg/ day thereafter. This regimen was chosen to achieve a plasma steady state sooner than 4 - 16 weeks that it takes on the standard dose of 20mg/ day. Although there are no published studies reporting the time steady state will be achieved with our exact loading dose regimen, a study of patients with metastatic breast cancer reported a loading dose schedule of 80mg/ day for 7 days followed by 20 mg/ day thereafter, allowed steady-state values to be reached in one week. Studies describing the pharmacokinetics of standard dose tamoxifen (10-30mg/ day), report steady state serum levels of 100ng/ml to 333ng/ml, levels sufficient to induce oesophageal adenocarcinoma cell growth arrest in vitro. The loading dose of tamoxifen and maintenance regimen proposed should be sufficient to observe the effect of cancer cell growth in vivo as the plasma steady state levels achievable with such dose are of sufficient concentration to inhibit oesophageal cell growth in the two in vitro studies.

A loading dose of 80mg/ day was chosen as it is the highest dose reported in the literature which isn't associated with an increased risk of serious adverse events. Tamoxifen has been used in infertility treatment for many years and is licenced for use in the UK for anovulatory infertility with doses of up to 80mg/ day for 4 consecutive days. Numerous studies report outcomes with doses of 20mg - 80mg/ day for 3 - 8 days, and no serious adverse events such of thromboembolism or stroke have been reported. In addition to infertility treatment, other studies of metastatic renal cell carcinoma (8 weeks), cervical cancer (5 days) and metastatic breast cancer (7 days) have reported outcomes with 80mg/ day and also do not report any serious adverse events. A period of 4 days was chosen for the loading dose regimen as it is already licensed for this duration in the UK and the majority of studies reporting the safety of 80mg/ day are for this time period. Having reviewed the literature, the investigators feel a loading dose regimen of 80mg/ day for 4 days is the highest safe dose which will allow a plasma steady state to be achieved as quickly as possible, allowing sufficient time to observe the biological effect of tamoxifen on oesophageal cancer, allowing valid conclusions to be made. The rationale for the loading dose regimen is to limit the time from recruitment (starting tamoxifen) to biopsy, ensuring patients are well enough to attend for the gastroscopy, as it is well known that this cohort of patents experience a deterioration in their quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients with oesophageal cancer who are not candidates for surgical resection or further chemotherapy.
* Men aged 18 - 95.
* Women aged 55 - 95.
* Patients who have a biopsy specimen of the cancer stored in the laboratory from the time of diagnosis.
* The patient agrees and is able to return to the same research facility for the gastroscopy.
* The patient has been informed of the nature of the study, agrees to its provisions, and has provided written informed consent as approved by the Institutional Review Board/Ethics Committee (IRB/EC) of the respective clinical site.

Exclusion Criteria:

* Chemotherapy within 4 weeks of entry into the trial.
* Life expectancy <4 weeks
* Concurrent hormonal therapy e.g. Any SERMs, Hormone Replacement Therapy, Oral Contraceptive, or within 4 weeks of entry into the trial.
* Concurrent anticoagulant therapy other than Aspirin.
* Concurrent aminoglutethimide, and droperidol drugs.
* Previous thromboembolic disease (DVT/ PE), stroke or transient-ischemic attack.
* A positive family history (first-degree relative) of confirmed idiopathic venous thromboembolic events (DVT/ PE).
* Bleeding diathesis or thrombocytopenia.
* Women of childbearing age/ pre-menopause (<55 years of age).
* Any other medical condition, which in the opinion of the investigator should be excluded from the study.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-12; Primary Completion 2018-08 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
A change in Ki67 expression following tamoxifen therapy, by comparing the pre- and post- tamoxifen biopsies | 1.5 years
  A change in Ki67 expression will be determined by immunohistochemistry on the specimens which will be fixed in formaldehyde and processed into paraffin blocks.

SECONDARY OUTCOMES:
A change in ER-α expression | 1.5 years
  A change in ER-α expression will be determined by immunohistochemistry on the specimens which will be fixed in formaldehyde and processed into paraffin blocks.
A change in ER-β expression | 1.5 years
  A change in ER-β expression will be determined by immunohistochemistry on the specimens which will be fixed in formaldehyde and processed into paraffin blocks.

CONTACTS AND LOCATIONS:
Overall Officials: Raheela Khan, Principal Investigator — University of Nottingham
Locations (2):
- United Kingdom (2):
  - Graduate Entry Medical School, University of Nottingham, Derby, Derbyshire
  - Royal Derby Hospital, Derby